CLINICAL TRIAL: NCT06991491
Title: Ivonescimab With GnP and SBRT in Patients With Metastatic Pancreatic Cancer (WGOG-PAN 004): an Open-label, Single-arm, Phase II Trial of First-line Multimodal Therapy With Spatial Tumor Immune Microenvironment Analysis
Brief Title: Ivonescimab With GnP and SBRT in Patients With Metastatic Pancreatic Cancer (WGOG-PAN 004)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Dan Cao, Chief physician, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025(352)
Record Dates: First submitted 2025-05-14; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GnP + Ivonescimab +SBRT (Experimental): Only one cohort of patients will be included, specifically those with pathologically confirmed metastatic pancreatic cancer and, who have not received any prior systemic anti-tumor therapy (including chemotherapy, radiation, or other investigational treatments) or those who have had prior radical pancreatic surgery for pancreatic cancer and have received regular postoperative adjuvant chemotherapy and have developed recurrence or metastasis more than 6 months after the last adjuvant chemotherapy.
  Interventions: Combination Product: GnP in combination with Ivonescimab and SBRT

INTERVENTIONS:
Combination Product: GnP in combination with Ivonescimab and SBRT — Gemcitabine 1000mg/m2, ivgtt,vdays 1 and 8, nab-Paclitaxel 125mg/m2, ivgtt, days 1 and 8 in combination with Ivonescimab 20mg/kg d1, every 21 days. Cycle 2 will be synchronized with primary or metastatic SBRT.

SUMMARY:
The aim of this study is to explore the efficacy and safety of a new combination regimen of GnP regimen, SBRT and the anti-PD-1/VEGF bis-antibody, Ivonescimab, in patients with recurrent metastatic advanced pancreatic cancer. The efficacy predictive biomarkers of this combination regimen will be further explored through information such as spatial analysis of the tumor immune microenvironment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed metastatic pancreatic cancer;
2. Patients who have not received any prior systemic anti-tumor therapy, or who have undergone prior radical pancreatic cancer surgery and received regular postoperative adjuvant chemotherapy, and who have developed recurrence or metastasis more than 6 months after final adjuvant chemotherapy;
3. Aged 18 to 75 years old;
4. Eastern Cooperative Oncology Group performance status score (ECOG) ≤ 2;
5. According to imaging and surgical evaluation, the liver lesion is unresectable or rhe patient is unable to tolerate surgery, and the primary lesion has no serious complications (perforation, obstruction or hemorrhea that cannot be managed by medical therapy);
6. At least one measurable tumor lesion: length and diameter of spiral CT greater than or equal to 10 mm, lymph node short diameter greater than or equal to 15 mm; maximum diameter of conventional CT or physical examination greater than or equal to 20mm;
7. Adequate organ functions as follows:

   Absolute neutrophil count ≥1500/mm3, leukocyte≥4000/mm3, platelet count ≥80,000/mm3, hemoglobin ≥9.0 g/dL; total bilirubin≤2.0 × upper limit of normal (UNL); serum creatinine ≤1.5 × UNL; alanine aminotransferase, aspartate aminotransferase ≤5 × UNL;
8. Life expectancy of longer than 3 months;
9. No history of autoimmune disease and no current co-morbid autoimmune disease;
10. Participate the study voluntarily and sign the informed consent document.

Exclusion Criteria:

1. Subjects with a known allergy to any of the study medications;
2. Subjects with known or suspected CNS metastases, i.e., subjects with signs or symptoms suggestive of the development of CNS metastases, unless CNS metastases have been ruled out by CT or MRI;
3. History of other malignancies within 5 years (except adequately treated basal cell carcinoma of the skin and carcinoma in situ of the cervix);
4. Anti-tumor therapeutic measures other than the treatment regimen of this study must be used concurrently during the study period, including chemotherapy, targeted therapy, hormone therapy, immunotherapy regimens, radiotherapy, and anti-tumor herbal treatments;
5. Prior use or ongoing use of chemotherapy, FAK inhibitor analogs, or anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4) antibodies;
6. Diagnosis of immunodeficiency or undergoing chronic systemic steroid therapy (administration of more than 10 mg of prednisone or equivalent per day) or any other form of immunosuppressive therapy within 7 days prior to administering the first dose of this study;
7. Patients receive live vaccines (including, but not limited to: measles, mumps, rubella, varicella/herpes zoster, yellow fever, rabies, BCG, and typhoid vaccines) within 30 days prior to their first dose of study drug therapy, and the use of virus-killed vaccines such as injectable seasonal influenza vaccine is permitted, but the use of live attenuated vaccines such as intranasal influenza vaccine (e.g., fluoride mist) is not permitted;
8. Uncontrollable hypertension (defined as systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg after treatment);
9. significant cardiac disease, including congestive heart failure (NYHA Class III-IV), previous myocardial infarction, or uncontrolled angina within 6 months;
10. Arrhythmia requiring treatment, including atrial fibrillation, supraventricular tachycardia, ventricular tachycardia, or ventricular fibrillation, with ECG abnormalities confirmed by review and in the judgment of the Investigator requiring clinical intervention or treatment;
11. History of a hemorrhagic or thromboembolic event within the last 6 months, e.g., cerebrovascular accident (including transient ischemic attack), pulmonary embolism, spontaneous hemorrhage from a tumor;
12. need for surgical intervention within 28 days or within 28 days of anticipated last dose
13. Combination of uncontrollable third cavity effusion, such as massive pleural effusion or ascites;
14. Previous gastrointestinal perforation or suspected gastrointestinal perforation;
15. Combinations of medications that, in the judgment of the investigator, must be used during the trial that may affect the metabolism of the product: e.g., strong CYP 3A4 inhibitors or inducers, primarily metabolized by CYP 3A4, 2C8, 2C9, 2C19, or 2D6, and medications with a low therapeutic index;
16. Persons with severe mental disorders;
17. Women who may be pregnant, gestating, or breastfeeding;
18. Subjects of childbearing age who are unwilling to use contraception during the trial period up to 3 months after the last dose;
19. Participation in a clinical trial of another drug or medical device within 4 weeks prior to the trial;
20. those who, in the judgment of the investigator, are not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
6-month-PFS rate | Follow up with patients for up to 24 months
  Proportion of patients with progression-free survival at 6 months.